CLINICAL TRIAL: NCT03678311
Title: Obstructive Sleep Apnea and Cardiac Electrophysiologic Biomarkers of Sudden Cardiac Death
Brief Title: Long QT Syndrome and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Reena Mehra, MD, Director, Sleep Disorders Research, Neurologic Institute, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1433
Record Dates: First submitted 2018-09-05; First posted 2018-09-19 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Long QT Syndrome; Sleep Apnea
MeSH Terms: conditions — Long QT Syndrome; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sleep Apnea ahi > 5 (Other): If Sleep Apnea index is > 5 and diagnosed with Long QT Syndrome
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — If diagnosed with Long QT Syndrome and have Sleep Apnea index >5 pauses per hour then given CPAP to wear for approximately 3 months.

SUMMARY:
Obstructive sleep apnea (OSA) has been associated with cardiac repolarization abnormalities and implicated in sudden cardiac death. A biologically plausible mechanism by which OSA exerts this lethality is by QT interval prolongation, a known marker of ventricular tachyarrhythmias (VTA) leading to cardiac death. Congenital long QT syndrome (LQTS) is a familial arrhythmogenic disorder characterized by prolonged QT interval on the electrocardiogram and increased propensity for VTA. Preliminary data identify an association of the extent of severity of OSA and progressive prolongation of the corrected QT interval in LQTS.

DETAILED DESCRIPTION:
Potential participants will come to the Cleveland Clinic Clinical Research Unit (CRU) for informed consent, eligible participants will undergo a 12 lead electrocardiogram. If the participants is found to have long QT syndrome (QTc ≥ 450 in men ad ≥ 470 in women) the participant will continue on in the study. If the participant is found to not have long QT syndrome the participant will exit the study. If continuing on in the study the participant will undergo a fasting venipuncture and blood pressure measurements. The participant will then be shown how to use the portable sleep study hook-up and continuous 12-lead ECG monitoring to be monitored in the home setting. The sleep study and ECG monitors will be returned by a courier service the next morning.

Those participants who are identified to have OSA (apnea hypopnea index>5, estimate 50% of those recruited) on the portable sleep monitoring will be invited to wear CPAP for 2-3 months with a follow up visit with repeat portable polysomnographic and continuous electrophysiologic assessments and CRU visit for bloodwork and blood pressure.

DATA COLLECTION Portable Polysomnography The Embletta Gold ® is a battery-operated device that can sample data at a 1000 Hz sampling rate and store data at 200 Hz, with 1 GB of storage capacity allowing storage of data from up to 20-24 hrs of recording. The device contains the critical sensors which are recommended by the American Academy of Sleep Medicine as validated sensors for measuring OSA: nasal pressure/flow; thoracic and abdominal inductance plethysmography (effort); and finger pulse oximetry (oxygen saturation).

Relevant PSG Variables: A registered polysomnologist will score the sleep study data. Apneas will be classified as "central" or "obstructive" according to the absence or presence of respiratory effort respectively. Hypopneas will be scored as a 50% amplitude reduction in inductance or flow and associated 3% oxygen desaturation or arousal. Periodic breathing will be defined as airflow or inductance channels increasing and decreasing at least 50% from the maximum, in a cyclic waxing and waning or "sinusoidal" manner for a consecutive period of >10 min.

Continuous Overnight 12-lead ECG Monitoring CardioDay Holter (GE) monitoring reads SEER 12 data and exports Holter data as individual 10 second, 12 lead reports up to six per minute, i.e. all recorded data. The monitor is capable of continuous 12-lead ECG monitoring with the ability to record up to 10 days with Bluetooth ® technology and 12-bit signal resolution with up to 1024 sampling rate.

ECG Sensor Application. This will be performed by a trained research coordinator at the visit in tandem with sleep monitor lead hook-up. Participants will be asked to remove clothing from the waist up to attach the sensors to the chest. Staff will ensure privacy by covering the participant with a sheet or gown. The staff will shave necessary areas on the chest prior to sensor application to ensure that the sensors stick closely to the skin and will provide the participant with the ECG monitor/holster/clip, leads, communicator and charger, electrodes and a handbook with simple pictorial/written educational instructions. A research coordinator will be available by phone 24-7 to address issues with device malfunction, lead placement and replacement of equipment. ECG quality grade data will be collected: (excellent: >90% of ECG data without artifact, good: 70-90% without artifact, fair: 50-70% without artifact, poor <50% artifact free).

Relevant ECG Variables. Standard average QT interval measures will be obtained with eventual ability to examine peri-apneic and peri-hypopneic alterations in QT interval. Novel QT morphologic assessments will be made with the GE compatible platform described below.

Novel QT analysis platform An analysis system which enables biopharmaceutical companies to analyze detailed morphology of the electrocardiography (ECG) T-wave (QT Guard Plus™, eResearchTechnology, Inc.). The system identifies and quantifies characteristic changes in the shape of the T-wave found in drugs that produce Torsades de Pointes (TdP), the latter a potentially lethal tachyarrhythmia. QT Guard Plus imports individual 10 second, 12 lead reports for analysis and parameter extraction, i.e. T wave shape measures with the capability to extract other electrophysiologic signatures as well.

Resting Blood Pressure BP will be measured after the participant has been sitting quietly for at least 5 minutes following standardized guidelines using a calibrated sphygmomanometer. Cuff size will be determined by measuring the circumference of the upper arm, measured at the midpoint and identifying the appropriate bladder size from a standard chart. Measurements will be repeated three times and recorded.

Fasting Venipuncture Phlebotomy (40cc) will be performed the morning of the baseline and follow-up visits using standard techniques by trained research staff following written procedures (e.g., pre-labeled bar coded tubes, minimizing trauma, etc.). The sample will be divided into tubes for the varied analyses (20 mL clot for serum, 20 mL EDTA). Clots will be centrifuged and the serum removed within 1 hr of venipuncture. Plasma from EDTA samples will be stored for future DNA analysis. Assays will be stored in dedicated, alarmed freezers at -80°C in the CRU Core Lab and transferred to designated space in the Pathology and Laboratory Medicine Institute.

Morning blood work to examine the association of electrolytes in relation to QT interval duration and stability upon follow up after use of CPAP. With collateral funding, bloodwork will allow for examination of markers of systemic inflammation which may serve as intermediary pathways for cardiac electrophysiologic biomarkers of VTA in OSA.

Continuous Positive Airway Pressure Intervention Participants randomized to CPAP will be provided with an Autopap REMstar device (Philips-Respironics, Inc, Murrysville, PA) with integrated humidifier, set at a pressure range of 4-20 cm H2O, with auto-titration according to the device's algorithm for detecting airflow limitation which provided wireless transmission of usage information to our research team.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of QT prolongation as described above
* Age 18-75 years
* Individuals able to participate in at least 2 overnight sleep and hysiologic assessments over a 3 month period.

Exclusion Criteria:

* Use of specific OSA treatments (CPAP, oral appliances)
* Use of supplemental oxygen
* Severe chronic insomnia
* Circadian rhythm disorder (e.g. shift work sleep disorder, delayed or advanced sleep phase syndrome)
* Insufficient sleep syndrome defined by reported sleep duration < 4 hours
* Unstable medical conditions (e.g., new onset or changing angina, a myocardial infarction or congestive heart failure exacerbation documented within the previous 3 months, uncontrolled hypertension (BP>170/110), uncontrolled diabetes mellitus (HbA1c>9.0), uncontrolled hypo- or hyperthyroidism)
* Psychiatric disorders which are inadequately treated
* Compromised competence
* Alcohol abuse (currently drinks >5 alcoholic drinks/day)
* Inability to provide informed consent
* Illicit drug use over last 6 months.

Rationale for criteria:

Patients with sleep disorders will be excluded as other sleep disorders may influence arrhythmogenesis.

Those on treatment for SDB will be excluded because treatment would preclude assessment of OSA pathophysiologic effects on QT biomarkers.

Those with unstable medical conditions or rapid or uncontrolled heart rate will be excluded due to safety reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reena Mehra, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available de-identified, non-sensitive, individual-level information on objective sleep characteristics, subjective sleep health and medical history (e.g. comorbid factors and medication use) and sociodemographics (e.g., age, gender education level). We will submit the data generated from the current proposal to the NIH funded National Sleep Research Resource (NSRR). The National Sleep Research Resource (NSRR) offers free web access to large collections of de-identified physiological signals and clinical data elements collected in well-characterized research cohorts and clinical trials. The NSRR is a public resource which provides opportunities for investigators to address critical scientific questions of interest.
Supporting Information: Study Protocol
Time Frame: When the study is complete.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was delayed in starting. Start Date 3/13/2019, End Date 4/30/2019. Recruited people with a clinical diagnosis of QT Prolongation that were not on treatment for sleep disordered breathing, chronic sleep disorders, unstable medical conditions or rapid/uncontrolled heart rate (for safety reasons).
Pre-assignment Details: Baseline Study 9 completed, 4 qualified to continue and receive CPAP. Zero started the 3 month follow up (CPAP treatment). Because of contract issues CPAPs were not available. Study ended 4/30/2019.
Period: Overall Study
Arm/Group | Sleep Apnea Ahi > 5
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Sleep Apnea index is > 5 and diagnosed with Long QT Syndrome
Arm/Group | Sleep Apnea Ahi > 5
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (4.8)
Apnea Hypopnea Index (AHI) [Median (Inter-Quartile Range); unit: events per hour] | 4.4 [3.5 to 9.4]
Percent of Sleep Time with SaO2<90% [Median (Inter-Quartile Range); unit: percent of sleep time] | 7 [0 to 19]
%SpO2 [Mean (Standard Deviation); unit: percent of oxygen saturation] | 99.1 (1.2)
STOPBANG [Mean (Standard Deviation); unit: units on a scale] — The STOPBANG questionnaire is a screening tool of obstructive sleep apnea. It sums up the number of events with range from 0 to 8, which include snoring, tiredness, observation of apnea, high blood pressure, high body mass index, age older than 50, large neck circumference and gender male. The higher STOPBANG score, the higher risk of obstructive sleep apnea.
  units on a scale | 3.2 (1.7)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions (0-3 for each). The total ESS score sums up 8 items with range 0-24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their daytime sleepiness.
  units on a scale | 9.9 (3.1)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is the depression module. It is a self-administered questionnaire with 9 questions (0-3 for each). The total PHQ-9 score sums up 9 items with range 0-27. The higher the PHQ-9 score, the higher severity of depression.
  units on a scale | 8.2 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: QT Interval (Corrected) Baseline Visit
Description: To examine the extent that OSA severity from overnight polysomnograph is associated with corrected QT interval (QTc) from daytime 12-lead ECG. The 24 hour continuous ECG is not available.
Time Frame: The 12-lead ECG will be collected in the morning and the overnight polysomnography will be the duration of their sleep for the night.
Measure: Mean (Standard Deviation); unit: square root of seconds
Arm/Group | Sleep Apnea Ahi > 5
Number analyzed (Participants) | 9
square root of seconds | 453.4 (28.7)
Statistical Analysis 1: Comparison: Sleep Apnea Ahi > 5; Spearman's correlation was used to evaluate the relationship between the outcome and the apnea hypopnea index; Test type: Other — The correlation between the outcome and AHI was tested by Spearman's correlation; p = 0.73, Spearman's correlation; Spearman's correlation = 0.13, 95% CI 2-sided [-0.75 to 1.00]

2. Primary Outcome: QT Interval (Corrected) Follow up Visit
Description: as for outcome 1
Time Frame: The 12-lead ECG will be collected in the morning and the overnight polysomnography will be the duration of their sleep for the night. This will be collected at their follow up visit after wearing CPAP for 2-3 months.
Population: No patient started follow up (3 Month CPAP Treatment). Because of contract issues CPAPs were not available.
Arm/Group | Sleep Apnea Ahi > 5
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of OSA Treatment on QTc
Description: To investigate the change in LQTS after OSA treatment with 2-3 month continuous positive airway pressure (CPAP) on QTc collected from daytime 12-lead ECG in those with LQTS.
Time Frame: After wearing CPAP for approximately 2-3 month the 12-lead ECG will be collected in the morning and the overnight polysomnography will be the duration of their sleep for the night.
Population: No patient started follow up (3 Month CPAP Treatment). Because of contract issues CPAPs were not available.
Arm/Group | Sleep Apnea Ahi > 5
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all participants during the 24 hour baseline/screening visit. Participants that qualified for CPAP were not given CPAP due to contract issues therefore, their participation was ended after the baseline/screening visit.
Description: Adverse events were collected on all participants during the 24 hour baseline/screening visit. Participants that qualified for CPAP were not given CPAP due to contract issues therefore, their participation was ended after the baseline/screening visit. There were no adverse events to report for this 24 hour period.
Groups:
- Sleep Apnea Ahi >5: Sleep Apnea Index >5 and diagnosed with Long QT Syndrome
Arm/Group | Sleep Apnea Ahi >5
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Due to factors beyond the investigators including delays in contracts within the one year scope of funding, the positive airway pressure intervention for this study could not be conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03678311/Prot_SAP_000.pdf